CLINICAL TRIAL: NCT04226261
Title: Prediction of Infection in Patients With Rheumatic Disease at High Risk of Infection
Brief Title: Next Generation Pathogen Sequencing for Prediction of Infection in Rheumatic Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NGPSPIRD
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma or serum samples collected but not required for clinical care will undergo next generation pathogen sequencing.
Oversight: Data Monitoring Committee: No

SUMMARY:
The majority of patients diagnosed with rheumatic disease, such as systemic lupus erythematosus, inflammatory myositis, and vasculitis, will experience fever or infection during their course of therapy. The most common microbiologically documented infection is bacterial, virus, and fungal, which can be associated with the severity and mortality of disease. Current methods of diagnosis require a significant load of pathogen making early detection difficult. Delayed diagnosis and delayed optimal therapy of infection are associated with increased morbidity and mortality.

This study seeks to identify whether next generation sequencing (NGS) of pathogens can identify patients with infection treated with corticosteroid and immunosuppressive agents. This would enable preemptive targeted therapy to replace prophylaxis treatment which often leads to some adverse events and antibiotic resistance.

DETAILED DESCRIPTION:
Plasma/Serum samples collected but not required for clinical care (discarded samples) will be collected and stored. Results of NGS will be compared between patients who develop definite infection immediately (within 72 hours) after sample collection, and those who remain well. Clinical data describing baseline information about the patient and rheumatic diseases, antibiotic and steroid or immunosuppressor therapy exposure, pathogen testing, immunology results, and infection-related events will be collected prospectively from the electronic medical record.

An initial exploratory phase will examine approximately 50 participants to determine whether the effectiveness of predicting infections. The study may then enroll up to 200 participants to collection additional data for analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 70 years;
* Undergoing care for rheumatic disease at Peking University People's Hospital;
* In a category of patients who are considered by the investigator to be at high risk of infection

Exclusion Criteria:

* Any condition that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who are being treated at Peking University People's Hospital and who have a high risk of infection.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-15 (Estimated); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of NGS-positive results | Once (within 72 hours of enrollment)
  To estimate the sensitivity of next generation pathogen sequencing for prediction of infection, the proportion of NGS-positive results in all positive infection will be given.
Proportion of NGS-negative results | Once (within 72 hours of enrollment)
  To estimate the specificity of next generation pathogen sequencing for prediction of infection, the proportion of NGS-negative results in all negative infection will be given.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, M.D, Ph.D, Principal Investigator — Peking University People's Hospital

REFERENCES:
- [Background] Goggin KP, Gonzalez-Pena V, Inaba Y, Allison KJ, Hong DK, Ahmed AA, Hollemon D, Natarajan S, Mahmud O, Kuenzinger W, Youssef S, Brenner A, Maron G, Choi J, Rubnitz JE, Sun Y, Tang L, Wolf J, Gawad C. Evaluation of Plasma Microbial Cell-Free DNA Sequencing to Predict Bloodstream Infection in Pediatric Patients With Relapsed or Refractory Cancer. JAMA Oncol. 2020 Apr 1;6(4):552-556. doi: 10.1001/jamaoncol.2019.4120. PMID 31855231
- See also: Next Generation Pathogen Sequencing for Prediction of Adverse Events — https://www.clinicaltrials.gov/ct2/show/NCT03226158?id=NCT02505568+OR+NCT02756650+OR+NCT01960790+OR+NCT02648581+OR+NCT02985775+OR+NCT04056533+OR+NCT01185223+OR+NCT03226158&draw=2&rank=2&load=cart